CLINICAL TRIAL: NCT00489840
Title: Treatment of Chronic Central Serous Chorioretinopathy With Open-label Anecortave Acetate
Acronym: CSC-AA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: LuEsther T. Mertz Retinal Research Center (Other); Alcon Research (Industry)
Responsible Party: Principal Investigator, Joan, Lawrence A. Yannuzzi, M.D., Manhattan Eye, Ear & Throat Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSC-AA
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Central Serous Chorioretinopathy
Keywords: Chronic Central Serous Chorioretinopathy
MeSH Terms: interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anecortave acetate (Experimental)
  Interventions: Drug: Anecortave Acetate Sterile suspension 15 mg; Drug: Anecortave Acetate

INTERVENTIONS:
Drug: Anecortave Acetate Sterile suspension 15 mg — anecortave acetate sterile suspension 15 mg., juxtascleral injection, every 6 months. for 24 months
  Other Names: retaane
Drug: Anecortave Acetate — anecortave acetate suspension 15 mg. juxtascleral injection every 6 months for 24 months.
  Other Names: retaane

SUMMARY:
Investigation to evaluate Anecortave Acetate in the treatment of chronic central serous chorioretinopathy

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is a disease of the macula characterized by loss of vision from exudation of fluid under the retina localized to the posterior pole. Acute central serous chorioretinopathy (CSC) has been defined as an idiopathic detachment of the neurosensory retina in the macular region associated with a focal leak at the level of the retinal pigment epithelium on fluorescein angiography. This area of leakage usually corresponds to a defect in retinal pigment epithelium (RPE). An acute episode of CSC usually resolves within 3 months from the time of onset with almost total restoration of the visual acuity.

However, in a more severe form of the disease, chronic central serous chorioretinopathy, there is diffuse decompensation of the RPE, recurrent retinal detachments, and progressive loss of visual acuity. Indocyanine green angiography shows diffuse hyperpermeability of the choriocapillaris layer. This chronic form of CSC is usually bilateral, and often causes severe vision loss and impaired quality of life for the patient. Chronic central serous chorioretinopathy can be defined on the basis of two factors: 1) persistence of the detachment for more than 6 months and 2) chronic recurrent acute detachments with widespread decompensation of the retinal pigment epithelium.

The standard of care for acute CSC is observation for a period of up to 3 months. If there is no complete resolution of the retinal detachment by 3 months, focal laser photocoagulation therapy may be used to treat the area of leakage. This treatment is usually effective in stopping leakage of fluid under the retina and causing resolution of the detachment. However, laser photocoagulation therapy is not beneficial in the treatment of chronic CSC because there is not a single easily identifiable point of leakage but rather diffuse disease of the RPE, thus rendering laser treatment ineffective. Because of the limitations of laser photocoagulation for chronic CSC, other treatments are currently under evaluation.

Corticosteroids appear to be intimately related to the pathogenesis of the disease. Exogenous corticosteroids have been shown to induce the disease via a variety of routes, whether oral, intravenous, intranasal, or intraarticular. Secondly, patients with endogenous hypercortisolism, such as those with Cushing's syndrome or with a type A personality, are also at increased risk of developing the disease.

The purpose of this medical research study is to evaluate Anecortave Acetate as an approach which may benefit patients with chronic CSC. Anecortave acetate is a novel agent, derived from the steroid cortisone, but modified to eliminate glucocorticoid effects via removal of the 11β-hydroxyl group, addition of a double bond at C9-11, and addition of an acetate group at C21 to increase ocular penetration and stability. Anecortave acetate has recently been shown to possess anti-glucocorticoid effects in the eye, such as in blocking steroid-induced glaucoma. Anecortave acetate treatment to the eye has been evaluated for other disorders, such as macular degneration, and boasts an outstanding safety record, with no adverse systemic reactions. Ocular adverse events were mild, such as subconjunctival hemorrhage.

The concept of this protocol is that if Anecortave Acetate blocks the steroid receptors for glaucoma and prevents steroid-induced glaucoma, perhaps it blocks the the steroid induced receptors involved in the pathogenesis of central serous chorioretinopathy. If successful, this modality of treatment may reduce the risk of progressive visual damage due to chronic CSC and perhaps even improve visual function without causing destruction to the overlying neurosensory retina.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female, of any race with clinical signs of chronic CSC:Evidence of chronic central serous chorioretinopathy and clinical/angiographic findings typical of the disease of greater than 6 months duration. Chronic central serous chorioretinopathy can be defined on the basis of two factors: 1) persistence of the detachment for more than 6 months and 2) chronic recurrent acute detachments with widespread decompensation of the retinal pigment epithelium
2. Patient must have best corrected ETDRS visual acuity between 20/40 and 20/320 in the Study Eye and visual acuity of 20/800 or better Fellow Eye
3. Patient must be willing, able to comply with the protocol, and provide informed consent.

Exclusion Criteria:

1. Patient with tears in retinal pigment epithelium.
2. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
3. Patients who have undergone intraocular surgery within last 2 months or capsulotomy within last month in study eye
4. Patient participating in any other investigational drug study.
5. Inability to obtain photographs to document CNV (including difficulty with venous access)
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to indocyanine green or iodine.
8. Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To investigate the use of Anecortave Acetate in patients with chronic central Chorioretinopathy | 24 months

SECONDARY OUTCOMES:
•Mean change in ETDRS Visual Acuity at 4 meters compared to baseline •Mean change in central retinal thickness as measured by OCT . -Change in leakage area seen during fluorescein angiography and ICG | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (2):
- United States (2):
  - Manhattan Eye, ear & Throat Institute, New York, New York
  - Vitreous-Retina-Macula Consultants of New York,PC, New York, New York